CLINICAL TRIAL: NCT07226453
Title: A Target Validation and Efficacy Study of Metformin in Patients With Recurrent or Progressive Posterior Fossa Group A (PFA) Ependymoma
Brief Title: Target Validation and Efficacy of Metformin in Patients With Posterior Fossa Group A (PFA) Ependymoma
Acronym: PNOC041
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The Lilabean Foundation, Inc. (Unknown); Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25087; NCI-2025-08332 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Posterior Fossa Ependymal Tumor
MeSH Terms: interventions — Metformin; Magnetic Resonance Spectroscopy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Target Validation (TV) Phase (Metformin) (Experimental): Participants will each receive daily oral metformin with a weekly schedule starting at 250 mg/m^2 twice a day (BID) for the first week, then increasing to 500 mg/m^2 BID for week 2, 1000 mg/m^2 BID for week 3, and then 1666 mg/m^2 BID for week 4-6 prior to planned surgery. Participants with no measurable disease following surgical intervention may either go off treatment or continue metformin at the physician's discretion. Participants have the option of continuing on the efficacy phase of the study without undergoing planned surgery no demonstrated progressive disease on pre-surgery MRI AND if the family opts to continue treatment with metformin without undergoing surgical resection of the tumor. Participants with measurable tumor by RAPNO criteria following surgery may continue onto efficacy phase and receive maintenance metformin until disease progression or till there are unacceptable adverse event(s).
  Interventions: Drug: Metformin; Procedure: Planned Surgical Resection; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Specimen Collection; Procedure: MR spectroscopy (MRS)
- Efficacy Phase (Metformin) (Experimental): Participants with recurrent or progressive PFA ependymoma that have failed upfront surgery and radiation will receive daily oral metformin until disease progression or till there are unacceptable adverse event(s). Disease response will be assessed by MRI imaging using RAPNO criteria. Participants already enrolled on the TV phase may enroll in this phase if they have measurable disease post-surgery. Treatment may continue until disease progression or until there are unacceptable adverse event(s).
  Interventions: Drug: Metformin; Procedure: Planned Surgical Resection; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Specimen Collection; Procedure: MR spectroscopy (MRS)

INTERVENTIONS:
Drug: Metformin — Given orally (PO)
  Other Names: Glucophage
Procedure: Planned Surgical Resection — Undergo planned surgery as part of regular care
  Other Names: Surgical Resection
Procedure: Magnetic Resonance Imaging (MRI) — Undergo MRI imaging
  Other Names: MRI
Procedure: Specimen Collection — Tumor Tissue, blood, and cerebral spinal fluid (CSF) may be collected for correlative analysis.
  Other Names: Specimen Sample Collection
Procedure: MR spectroscopy (MRS) — Undergo MRS imaging
  Other Names: MRS

SUMMARY:
This is a multi-site study of the pharmacodynamic effects and efficacy of metformin in children and young adults with recurrent or progressive Posterior Fossa Group A (PFA) ependymoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess pharmacodynamic effect on PFA tumor cells of metformin in participants with recurrent or progressive PFA undergoing surgical resection of the tumor by determining change in H3K27me3 and/or EZHIP expression in tumor nuclei compared to pre-treatment levels (TV Phase)

II. To measure disease stabilization rate by Response Assessment in Pediatric Neuro-Oncology (RAPNO) criteria (complete (CR), partial (PR) response; ≥50% reduction in size but <CR), and Stable (SD); < 50% reduction in size but not meeting criteria for progressive disease) in participants with recurrent or progressive PFA ependymoma following metformin treatment (Efficacy Phase).

EXPLORATORY OBJECTIVES:

I. Estimate the 1-year progression-free survival and overall-survival of participants with recurrent or progressive PFA treated with single agent metformin (Efficacy Phase).

II. To assess pharmacokinetics (PK) of metformin by measuring plasma, CSF and intra-tumoral concentration of metformin, the latter two obtained at the time of surgery or at the time of further disease progression on study in consenting participants (Both cohorts).

III. Evaluate the feasibility of using MR spectroscopy (MRS) imaging to study oncometabolite profile of recurrent or progressive PFA ependymoma pre-and post-treatment with metformin.

OUTLINE:

This will be a two-part study: a TV phase and an efficacy phase. Participants will be initially enrolled in the TV phase and receive treatment prior to planned surgery. Participants already enrolled on the TV phase may continue to the efficacy phase of the study if they have measurable disease post-surgery. Participants in the efficacy phase will receive daily oral metformin until disease progression or till there are unacceptable adverse event(s). Long term/survival follow-up procedures are to be captured under the Pediatric Neuro-Oncology Consortium (PNOC) Protocol for Children and Young Adults Diagnosed with a Central Nervous System (CNS) Tumor to Assess Cognitive, Quality of Life (QOL), and Comprehensive Effects of Therapies protocol (COMP). Participants will be followed under the PNOC COMP protocol until death or withdrawal from study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have recurrent or progressive posterior fossa A (PFA) ependymoma following surgery AND radiation treatment (RT).
2. Participants must have a diagnosis of PFA ependymoma either at initial diagnosis or at recurrence. Any number of previous recurrences are permissible provided the participant meets other enrollment criteria.
3. Participants must have adequate tumor tissue available from initial diagnosis or from pre- trial enrollment. Formalin-fixed paraffin-embedded (FFPE) material (1 full block) should be provided. If FFPE material is not available, 10 unstained slides with an accompanying hematoxylin and eosin (H&E) report should be provided.

   Target Validation (TV) Phase:

   o Participants are candidates to undergo elective surgery for removal of all or a portion of their recurrent/progressive tumor.

   Efficacy Phase:
   * Participant must have measurable disease; this will be defined as lesions that can be accurately measured in two dimensions (longest diameter to be recorded) The size threshold is met if both in-plane diameters are ≥10 mm or both in-plane diameters are at least two times the MRI slice thickness, plus the interslice gap with a minimum size of no less than double the slice thickness on MRI.
   * Participants with an isolated local progression of the tumor following RT (or stereotactic radiosurgery, SRS) must be > 6 months from completion of RT to the lesion to rule out pseudo progression or must have tissue confirmation of progression prior to enrollment.
   * Previously irradiated lesions are considered non-measurable except in cases of documented progression of the lesion since the completion of radiation therapy.
4. Prior Therapy: Participants must not be receiving metformin for other medical indications or previous exposure to metformin following their diagnosis of PFA ependymoma. However, participants treated on the TV phase, but did not continue onto maintenance therapy will be allowed to enroll on the efficacy phase with future recurrences or progression of their disease.
5. Age: 1 -39 years at the time of enrollment.
6. Performance Score: Karnofsky >= 50 for participants > 16 years of age and Lansky >=50 for participants <=16 years of age. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
7. Corticosteroids: Participants who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration.
8. Organ Function Requirements

   1. Peripheral absolute neutrophil count (ANC) >= 1000/mm^3.
   2. Platelet count >=100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
   3. Serum creatinine < 1.5 Upper Limit normal (ULN) based on age and gender
   4. Total bilirubin <= 1.5 x ULN for age; in presence of Gilbert's syndrome, total bilirubin < 3 x ULN or direct bilirubin < 1.5 x ULN
   5. alanine aminotransferase (ALT) <= 3 x ULN.
   6. aspartate aminotransferase (AST) <=3 x ULN.
9. Participants with seizure disorder may be enrolled if well controlled and are on stable dose of anti-seizure medication for > 72 hours prior to enrollment. Participants who have neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration.
10. Participants must enroll on PNOC COMP if PNOC COMP is open to accrual at the enrolling institution.
11. A legal parent/guardian or participant must be able to understand, and willing to sign, a written informed consent and assent document, as appropriate.

Exclusion Criteria:

1. Participants with a history of diabetes mellitus or those found to have pre-diabetes on HbA1C screening test are excluded from the study.
2. Participants without any measurable disease but with only isolated leptomeningeal disease progression.
3. Participants who have had chemotherapy or have received radiotherapy to the non-target lesion within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
4. Participants must be at least 7 days since the completion of therapy with a biologic or small molecule agent. For any agent with known adverse events that can occur beyond 7 days after administration, the period prior to enrollment must be beyond the time during which adverse events are known to occur. Such participants should also be discussed with study chairs.
5. Participants with rapidly progressive symptoms that require urgent surgery that in the investigators assessment cannot be safely deferred for 6 weeks are excluded from target validation phase of the study
6. Participants who are receiving any other investigational agents.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
9. Women of childbearing potential must not be pregnant or breast-feeding.
10. Human immunodeficiency virus- (HIV) positive participants will be ineligible if HIV therapy regimen has not been stable for at least 4 weeks or there is intent to change the regimen within 8 weeks following enrollment, or if they are severely immunocompromised.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with changes in biomarkers between the pre-and post-metformin treated samples (Target Validation Phase) | From initiation of study treatment until surgical resection of tumor, approximated 6 weeks
  Proportion of participants with a 10% reduction in Enhancer of Zeste Inhibitory Protein (EZHIP) and/or a 10% increase in the epigenetic modification to the DNA packaging protein histone H3, with tri-methylation of lysine 27 on histone H3 (H3K27me3) between the pre- and post-metformin treated samples by Immunohistochemistry (IHC).
Disease Stabilization Rate (Efficacy Phase) | From initiation of study treatment until discontinuation of treatment, up to 2 years
  The primary endpoint of the efficacy phase is the disease stabilization rate by RAPNO criteria (complete (CR), partial (PR); response >50% reduction in size < CR, and stable (SD) which is a < 50% reduction in size and not meeting the definition for progressive disease) tumor responses), CR+PR+SD.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, Principal Investigator — University of California, San Francisco; Santhosh A Upadhyaya, MD, Study Chair — University of Michigan, C. S. Mott Children's Hospital
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets may be shared with research collaborators during the course of the study.
Supporting Information: Study Protocol, SAP, ICF